CLINICAL TRIAL: NCT04611958
Title: Intraductal Liposomal Bupivacaine as a Therapeutic Trial to Determine the Contribution of Peripheral Versus Central Sensitization in the Pathogenesis of Pain in Chronic Pancreatitis- a Pilot and Feasibility Study
Brief Title: Intraductal Liposomal Bupivacaine for Chronic Pancreatitis
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The FDA requirements for the IND are not feasible to complete.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00268695
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bupivacaine arm (Experimental): Participants undergoing ERCP as part of routine clinical care will be consented for this study.
  Interventions: Drug: ERCP with Bupivacaine infusion

INTERVENTIONS:
Drug: ERCP with Bupivacaine infusion — Selective cannulation of the pancreatic duct with ERCP scope will be performed. Any contrast dye used will be carefully aspirated and the duct will be flushed with saline as necessary to clear all residual dye. The canula will be taken to the tail of the pancreatic duct, and gradually withdrawn with slow infusion of the bupivacaine solution. Liposomal bupivacaine (13.3 mg/ml of Exparel) will be injected into the main pancreatic duct for a total of 5-10 ml (depending on the length of the pancreatic duct).
  Immediately after the procedure, the patient will be monitored for any evidence of acute pancreatitis (worsening abdominal pain, with amylase or lipase x3 upper limit of normal). The patient will be questioned daily after the procedure for common side effects of bupivacaine including nausea, fever, change in taste, dizziness, weakness, palpitations and loss of taste or any other new or unusual symptom.

SUMMARY:
The major clinical features of chronic pancreatitis include glandular (exocrine and endocrine) failure and pain. Pain has remained a major clinical challenge and is present in up to 90% of patients and is the primary cause of hospitalization in most patients. Unfortunately, pain in chronic pancreatitis has been very difficult to treat.

The investigators hypothesize that the best method to reliably abolish peripheral nerve signaling is the use of a local anesthetic within the target organ (i.e. pancreas). This can best be done during endoscopic retrograde cholangiopancreatography (ERCP).

Since ERCP is done under deep sedation or general anesthesia, it is critical to select a local anesthetic whose effect persists well after recovery from the procedure; if not, the assessment of the effect of the local anesthetic on pain will be impossible to assess. The investigators have therefore chosen liposomal bupivacaine (Exparel, Pacira Pharmaceuticals), which is an FDA approved product for local infiltration that has a longer duration of action (up to 72 hours) and a slower absorption into the systemic circulation, avoiding high plasma concentrations.

DETAILED DESCRIPTION:
The major clinical features of chronic pancreatitis include glandular (exocrine and endocrine) failure and pain. The former can usually be managed satisfactorily by replacement strategies (enzymes or insulin) to restore nutritional and metabolic stability. However, pain has remained a major clinical challenge and is present in up to 90% of patients and is the primary cause of hospitalization in most patients. Unfortunately, pain in chronic pancreatitis has been very difficult to treat, and the investigators' lack of understanding about the underlying biology has led to various empirical approaches that are often based on purely anatomical grounds, and are generally highly invasive. Significant tissue injury such as that observed in chronic pancreatitis not only triggers nociceptor activation but over time, can also increase the pain in the whole system, a process called sensitization.

Determination of the contribution of peripheral versus central factors to nociceptive sensitization has significant clinical implications in an individual patient. Thus, if pain is caused primarily by signals emanating in the peripheral nerves, then perhaps invasive procedures directed against the pancreas (including pancreatectomy) are justified and can be expected to have a high probability of success. On the other hand, if central sensitization is the dominant pathophysiological factor, then these procedures may cause more harm than good and the patient may be best served using aggressive neuromodulator therapies.

The most direct way to address this question is to interrupt peripheral nerve signaling and determine how much of the pain, if any, is taken away. Unfortunately, there are no satisfactory methods to do this currently. Although celiac or splanchnic nerve blocks have been used for the treatment of pain in chronic pancreatitis, the treatments have had limited success for a variety of reasons, including the fact that the technique may not always be accurate in terms of the site of injection.

The investigators hypothesize that the best method to reliably abolish peripheral nerve signaling is the use of a local anesthetic within the target organ (i.e. pancreas). This can best be done during endoscopic retrograde cholangiopancreatography (ERCP), a technique in which the main pancreatic duct is cannulated with the help of a duodenoscope and contrast material injected. This technique is routinely done to assess pancreatic duct anatomy prior to consideration of a therapeutic intervention such as a stent, stricture dilation, or stone removal/lithotripsy.

Since ERCP is done under deep sedation or general anesthesia, it is critical to select a local anesthetic whose effect persists well after recovery from the procedure; if not, the assessment of the effect of the local anesthetic on pain will be impossible to assess. The investigators have therefore chosen liposomal bupivacaine (Exparel, Pacira Pharmaceuticals), which is an FDA approved product for local infiltration that has a longer duration of action (up to 72 hours) and a slower absorption into the systemic circulation, avoiding high plasma concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent
* Age >18 years
* Patients with an established diagnosis of chronic pancreatitis with constant daily pain consistent with the same and not relieved despite standard clinical care for at least 6 months and in whom ERCP is indicated for standard of care.

Exclusion Criteria:

* Significant liver or renal dysfunction.
* Any Contraindication of ERCP.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in the pain score at 24 hours after ERCP | 24 hours after the ERCP
  Raw pain score using a visual analog scale from 0 to 10, being 0 no pain and 10 the worst pain the participant can imagine.

SECONDARY OUTCOMES:
Change in the pain score at 2 hours after ERCP | 2 hours after ERCP
  Raw pain score using a visual analog scale from 0 to 10, being 0 no pain and 10 the worst pain the participant can imagine.
Change in the pain score at 48 hours after ERCP | 48 hours after ERCP
  Raw pain score using a visual analog scale from 0 to 10, being 0 no pain and 10 the worst pain the participant can imagine.
Change in the pain score at 72 hours after ERCP | 72 hours after ERCP
  Raw pain score using a visual analog scale from 0 to 10, being 0 no pain and 10 the worst pain the participant can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Pasricha, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hopital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No